

## **Consent Form**

Title of Research Study: Inflammation in infective endocarditis

Principal Investigator: Dr Daniel Harding, d.harding@qmul.ac.uk

IRAS Number: 353031

Thank you for your interest in this research.

Should you wish to participate in the study, please consider the following statements. Before signing the consent form, you should initial all or any of the statements that you agree with. Your signature confirms that you are willing to participate in this research, however you are reminded that you are free to withdraw your participation at any time.

| Statement | Please initial box |
|---|---|
| 1. I confirm that I have read the Participant Information Sheet dated [18_12_24] version [V1] for the above study; or it has been read to me. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| 2. I understand that my participation is voluntary and that I am free to stop taking part in the study at any time without giving any reason and without my rights being affected. | |
| 3. I understand that my data generated in this study will be accessed by the chief investigator and the clinical research team. | |
| 4. I understand that blood and heart valve samples will be collected from me (heart valve only if I undergo essential endocarditis surgery). | |
| 5. I understand that samples collected for this study will be moved and stored in the Chief Investigator's lab at Queen Mary University | |
| 6. I understand that the researcher will not identify me in any publications and other study outputs using personal information obtained from this study. | |

| 7. I agree to be conta | | | |
|---|---|---|---|
| 8. I agree to receivin | | | |
| I agree to my tissue samples being stored for subsequent studies in infective endocarditis. | | | |
| Optional Clauses | | | |
| Statement | | | Please initial box |
| 1. (If appropriate) I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | |
| 2. (If appropriate) I agree to my General Practitioner being informed of my participation in the study. | | | |
| important information<br>Queen Mary's Privac | about your persor<br>by Notice will be<br>tact Data Protection | privacy notice for research partice all data and your rights in this reprovided. If you have any queston Officer, Queens' Building, Mile Ed 20 7882 7596. | spect. A hard copy of<br>tions relating to data |
| Participant name | Date | Signature | |
| Name of person taking consent | Date | Signature | |
| I,any foreseeable risks a copy of this form. | | hat I have carefully explained the of the proposed research to the pa | |